CLINICAL TRIAL: NCT04535882
Title: Association Between Serum Leucine-rich Alpha-2 Glycoprotein Levels and Endoscopic Activity of Possible Ulcerative Colitis or Crohn's Disease Colitis
Brief Title: Effectiveness of Serum Leucine-rich Alpha-2 Glycoprotein Levels on IBD
Status: Completed | Type: Observational
Sponsor: Showa Inan General Hospital (Other)
Responsible Party: Principal Investigator, Akira Horiuchi, Chief, Showa Inan General Hospital
Other Study IDs: LRG
Record Dates: First submitted 2020-08-28; First posted 2020-09-02 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: LRG Levels

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: serum leucine-rich alpha-2 glycoprotein (LRG) levels — Patients who were diagnosed with possible UC or Crohn disease according to endoscopic, radiological, histological, and clinical criteria were enrolled. Serum samples were collected from patients, and scores for clinical and endoscopic activity of disease were obtained by reviewing the clinical records of patients. Serum sampling and colonoscopy were performed within 7 days.

SUMMARY:
We attempt to examine the association between serum leucine-rich alpha-2 glycoprotein (LRG) levels and endoscopic activity in patients with possible ulcerative colitis (UC) or Crohn's disease (CD) to determine whether LRG was a predicting marker for UC or CD.

DETAILED DESCRIPTION:
Serum samples were collected from patients, and scores for clinical and endoscopic activity of disease were obtained by reviewing the clinical records of patients. Serum sampling and colonoscopy with histology were performed within 7 days.The disease activity of UC and CD patients was evaluated by the Mayo score and Crohn disease activity index (CDAI), respectively. The Mayo endoscopy score was evaluated. UC patients whose Mayo endoscopy score was 2 or 3 were divided into the active UC group.

CD patients whose CDAI >150 were divided into the active CD group.

ELIGIBILITY:
Inclusion Criteria:

* Patients whom possible UC or Crohn disease was suspected

Exclusion Criteria:

* other autoimmune diseases
* acute or chronic renal failure
* chronic heart diseases
* liver cirrhosis
* cancer
* acute or chronic infections
* ischemic colitis
* infectious colitis

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: In total, a consecutive cohort of 300 patients with possible UC or CD will be enrolled in this study at our hospital.
Sampling Method: Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Serum LRG measurement | one year
  Serum samples were collected from patients, and scores for clinical and endoscopic activity of disease were obtained by reviewing the clinical records of patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Showa Inan General Hospital, Komagane, Nagano, Japan